CLINICAL TRIAL: NCT01298414
Title: Pediatric Myeloid Leukemia-Specific miRNA Expression Profiles Induced by the Leukemic Stem Cell Niche
Brief Title: Biomarkers in Bone Marrow Samples From Young Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML11B9; COG-AAML11B9 (Other: Children's Oncology Group); NCI-2011-02849 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AAML11B9 (Other: Children's Oncology Group)
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: childhood acute myeloid leukemia/other myeloid malignancies
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Bone Marrow
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: RNA analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of bone marrow from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer.

PURPOSE: This research study is looking at biomarkers in bone marrow samples from young patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To study the effect of niche mesenchymal stromal cells (MSC) exposure on microRNAs (miR) expression in pediatric AML at different time points and compare those profiles to the miR profiles at baseline.
* To focus on four pediatric AML-specific miRs (miR34a, miR538e, miR193e, and miR198) which show the most significant differential expression after in vivo niche exposure at four months (hematogenous spread).
* To determine whether altered miR expression reflects or causes the metastatic invasion pattern of AML.

OUTLINE: Bone marrow-derived mesenchymal stromal cell (MSC) samples are implanted subcutaneously in NOD/SCID mice. Cells are then harvested at day 0, 1 month, and 4 months post-implantation. miRNA is isolated and analyzed by Ilumina MicroRNA Expression Profiling single Beadchip. The obtained data is then analyzed by the Illumina Genome Studio Analysis Software.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia
* Fresh human bone marrow samples obtained from orthopedic surgery at the Tissue Donation Program of The Feinstein Institute and the Children Oncology Group (COG) Myeloid Disease Biorepository

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Diagnosis of acute myeloid leukemia
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
miR expression patterns in pediatric AML are regulated by the niche MSC-associated microenvironment
Exposure of AML cells to the niche MSCs generate changes in pediatric AML miR expression profiles
Correlation between changes in pediatric AML miR expression profiles and changes in biological behavior of AML cells (dormant versus invasive)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah R.I. Vaiselbuh, MD, Principal Investigator — Feinstein Institute for Medical Research